CLINICAL TRIAL: NCT02639858
Title: A Phase II Study to Evaluate the Efficacy and Safety of Docetaxel-PM in Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Study to Evaluate the Efficacy and Safety of Docetaxel Polymeric Micelle (PM) in Recurrent or Metastatic HNSCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOCH&N201
Record Dates: First submitted 2015-12-14; First posted 2015-12-28 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Docetaxel-PM (Experimental): Docetaxel-PM 75mg/m2 IV infusion
  Interventions: Drug: Docetaxel-PM

INTERVENTIONS:
Drug: Docetaxel-PM — Docetaxel PM 75mg/m2 IV infusion
  Other Names: Nanoxel M

SUMMARY:
A phase II study to evaluate the efficacy and safety of Docetaxel-PM in recurrent or metastatic head and neck squamous cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were histologically or cytologically diagnosed as having oral cavity, oropharynx, hypopharynx, or larynx squamous cell carcinoma with recurrent and metastatic evidence and who cannot be treated by salvage surgery or radiotherapy
2. Time of disease progression, regardless of whether that treatment or after platinum-based therapy

   ①Patients who have disease progression after concurrent chemoradiotherapy of curative purpose (including induction chemotherapy) including a platinum-based (cisplatin or carboplatin) chemotherapy

   ② Patients who have disease progression after primary or secondary treatment of palliative purpose including a platinum-based (cisplatin or carboplatin) chemotherapy
3. Patients who aged 20 years or older and under 79 years old
4. Patients whose Eastern Cooperative Oncology Group (ECOG) performance scores are 0-2
5. Patients who have one measurable lesion at least by RECIST criteria 1.1
6. Patients who show adequate function of organ:

   * bone marrow: Absolute Neutrophil count (ANC) ≥ 1,500/μL, Platelet count ≥ 100,000/μ, Hb≥ 9.0 g/dl (allowed blood transfusion)
   * Liver: ① with no evidence of liver metastasis; Total bilirubin ≤ 1.5mg/dl, alkaline phosphatase (ALP), aspartate transaminase (AST), alanine transaminase (ALT) ≤ 2.0 X upper limit of normal (ULN)

     ② with liver metastasis; bilirubin ≤ 3.0 X ULN, aspartate transaminase (AST), alanine transaminase (ALT) ≤ 5.0 X ULN
   * Kidney: creatinine ≤ 1.5 X ULN
7. Patients who have signed written consent forms prior to participation in the clinical trial

Exclusion Criteria:

1. Patients who have Primary tumor of nasopharynx
2. Patients who have received treatment prior regimen of three or more drugs
3. Patients who have Primary malignant tumors of other sites (except if; early cervical cancer, skin basal cell cancer received appropriate treatment, Malignant tumor without recurrent state treated five years previously)
4. Previous radiotherapy is allowed, patients who should be completed radiotherapy before 4 weeks prior to the initial administration of the investigational product
5. Patients who have received a major surgery within 4 weeks prior to the initial administration of the investigational product or patients who does not recover after major surgery
6. Patients who have severe diseases or medical condition as follows

   * Congestive heart failure(NYHA class III or IV)
   * Unstable angina, cardiac infarction within 6 months
   * Second-degree atrioventricular (AV) block or more, clinically cardiac arrhythmia that needs drug therapy
   * Uncontrollable Hypertension
   * Hepatic cirrhosis (≥ Child class B)
   * Interstitial lung disease
   * Mental disorder not to comply with the protocol
   * Uncontrolled diabetes
   * Uncontrolled ascites or pulmonary edema
   * Active infection
7. Pregnant or lactating women
8. Patients considered inappropriate to participating the study by the investigator

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2015-10; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Response rate as assessed by RECIST v1.1 | 2 years
  Response is confirmed at least 4 weeks later. Assessment: every 6 weeks (treatment period), every 2 months (follow-up period)

SECONDARY OUTCOMES:
Progression free survival (PFS) | 2 years
  Assessment: every 2 months (follow-up period)
Disease control rate (DCR) | 2 years
  DCR is defined as the percentage of patients who have achieved complete response, partial response and stable disease
Overall survival | 2 years
  Assessment: every 2 months (follow-up period)
Number of participants with adverse events as assessed by CTCAE v4.0 | 2 years
Incidence rate of hypersensitivity reaction to Docetaxel-PM | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Samyang Biopharmaceuticals, Seoul, South Korea